CLINICAL TRIAL: NCT00587587
Title: A Prospective, Randomized, Controlled Pilot Study of Apligraf for the Treatment and Prevention of Recurrence of Excised Keloids
Brief Title: A Pilot Study of Apligraf for the Treatment and Prevention of Recurrence of Excised Keloids
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Katherine B. Giovino, Director of Clinical Operations, Organogenesis Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-KEL-001-AG
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Apligraf (bilayered living cell therapy)
  Interventions: Device: Apligraf
- B (Active Comparator): Dressing regimen comprised of a primary nonadherent dressing, dry gauze dressing and bolster gauze dressing, if necessary
  Interventions: Other: Standard dressing regimen

INTERVENTIONS:
Device: Apligraf — Application at Day 0, potential re-application at Week 4
  Arms: A
Other: Standard dressing regimen — A primary nonadherent dressing, dry gauze dressing and bolster gauze dressing if necessary
  Arms: B

SUMMARY:
This pilot study will assess the safety and efficacy of Apligraf in the healing and recurrence of keloids post surgical shave excision in patients with clinically diagnosed keloids.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 65 years of age.
* Subject or legal guardian has read, understood, and signed appropriate Institutional Review Board (IRB) approved informed consent, photography release form and HIPAA consent in their own language.
* Subject with 1 keloid measuring between 1 cm2 - 40 cm2 as assessed by the Investigator, present for at least 6 months and a Beausang Scar scale combined score of 5 or greater.
* Subject is a male or female who must have a documented negative urine pregnancy test if of child bearing potential. Sexually active females must be practicing a medically proven form of contraception during the course of the study period.
* Subject and/or legal guardian must be able and willing to follow study procedures and instructions.
* Subject and/or legal guardian must be able and willing to return for follow-up study visits.
* Subject agrees to not use a keloid medication or injection treatment for four weeks prior to Day 0.
* Subject agrees not to use any other keloid treatments for the duration of the study.
* Subject is otherwise healthy as assessed and determined by the Investigator

Exclusion Criteria:

* Subject is suffering from a condition likely to require medical attention, including administration of any treatment which in the opinion of the Investigator could influence the results of the study.
* Subject with any systemic condition like uncontrolled diabetes mellitus (glycosylated hemoglobin, HbA1C > 10%), cancer (biopsy confirming active malignancy), positive HIV test, or any disorder(s) that may compromise wound healing.
* Subject is suffering from an abnormal skin condition on the affected area not usually associated with keloids such as psoriasis, or eczema.
* Subject who is currently or has received topical or systemic steroid medication therapy within the past four weeks affecting the course of the keloid and/or its evaluability. Inhaled steroid therapy is acceptable.
* Subject with the presence of acute infections in the areas intended for treatment.
* Subject with known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.
* Subject who is lactating or pregnant (positive result as determined by urine testing).
* Subject with liver (ALT/SGPT, ALP, AST/SGOT, bilirubin, albumin, total protein, LDH) and/or renal function (BUN and creatinine) tests > 2 x upper limit of normal (ULN).
* Subject who has been previously enrolled in any wound or investigational device study for any disease within the past four weeks.
* Subject who has received an investigational drug or biological treatment within the past three months.
* Subject previously treated with Apligraf, Dermagraft or any other cell therapy at the target keloid site.
* Subject with a history of alcohol or substance abuse within the previous year, which could interfere with study compliance such as inability to attend scheduled study visits or compliance with home dressing changes.
* Subject with a history of anaphylaxis.
* Subject who, in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Woolery-Lloyd, MD, Principal Investigator — University of Miami, Miller School of Medicine, Division of Cosmetic Dermatology; Damien Bates, MD, PhD, FRACS (Plast.), Study Director — Organogenesis Inc.
Locations (1):
- University of Miami, Miller School of Medicine, Division of Cosmetic Dermatology, Miami Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Apligraf: Apligraf (bilayered living cellular construct) plus a dressing regimen comprised of a primary nonadherent dressing, dry gauze dressing and bolster gauze dressing, if necessary
- Control: Dressing regimen comprised of a primary nonadherent dressing, dry gauze dressing and bolster gauze dressing, if necessary
Period: Overall Study
Arm/Group | Apligraf | Control
Started | 17 | 13
Completed | 11 | 12
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apligraf | Control | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 30
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.7 (12.9) | 36.7 (13.5) | 34.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 12 | 28
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Purpose of This Study Will be to Gain Preliminary Safety Experience With Apligraf in the Keloid Indication. The Number of Participants Experiencing AEs is Presented.
Description: Summary of all reported adverse events (AE) in the intent to treat (ITT) population.
  AE was defined as any adverse change in the subject's medical status compared with the subject's baseline condition, whether or not the event was related to the study device or a study procedure; or an exacerbation (either in frequency or severity) in a subject's pre-existing condition. AE data were collected at every study visit or if volunteered by the subject at any time during the study.
Time Frame: 52 weeks
Population: ITT analysis per protocol. Report of at least 1 treatment emergent AE.
Measure: Number; unit: Participants
Groups:
- A (Apligraf): Apligraf (bilayered living cell therapy)
- B (Control): Dressing regimen comprised of a primary nonadherent dressing, dry gauze dressing and bolster gauze dressing, if necessary
Arm/Group | A (Apligraf) | B (Control)
Number analyzed (Participants) | 17 | 13
Participants
  Any AE | 12 | 10
  Serious Adverse Event (SAE) | 0 | 0
  Unanticipated Adverse Device Effect (UADE) | 0 | 0
  Deaths | 0 | 0
Statistical Analysis 1: Comparison: A (Apligraf) vs B (Control); Fisher's exact test used to evaluate treatment differences between Apligraf subjects and Control subjects experiencing any AEs; Test type: Superiority or Other; p = 1.0000, Fisher Exact — P-value compares overall incidence of AEs between groups, ie Apligraf 12/17 and Control 10/13. UADE is defined in 21CFR812.3(s)

2. Secondary Outcome: Change in Degree of Keloid Recurrence as Measured by Beausang Scar Scale (BSS)
Description: Change in BSS cumulative score, Baseline to Last Visit, as reported by the Investigator, is reported.
  BSS is a composite score where the individual scores from the following categories are summed:
  Color (rated 1[perfect]-4[gross mismatch]), Shine (1/Matte or 2/Shiny), Contour (rated 1[flush with surrounding skin]-4[keloid]), Distortion (rated 1[None]-4[severe]), Texture (rated 1[normal]-4[hard]), and Overall Assessment on a 10cm visual analog scale (rated 0[excellent scar]-10 [poor scar]).
  Total score ranges from 5 (clinically well healed scar) - 28 (clinically poor scar).
Time Frame: Baseline to Week 52 or Last Visit
Population: Modified ITT (mITT) for randomized subjects only. Last Visit is the score recorded at last subject visit with non-missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
Units on a scale | -8.8 (5.1) | -9.7 (4.3)
Statistical Analysis 1: Comparison: Apligraf vs Control; Test type: Superiority or Other; p = 0.5863, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Cumulative Incidence of Keloid Recurrence at Week 52
Description: Recurrence is defined the first study visit at which the Investigator scores the Contour component of the BSS with a 4 (indicating a keloid). Contour is one of the five components measured in the BSS with Contour scores ranging from 1 (flush with surrounding skin) to 4 (keloid). Recurrence is a negative outcome.
Time Frame: 52 weeks
Population: Cumulative assessment, mITT population for randomized subjects only
Measure: Number; unit: participants
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
participants | 4 | 2
Statistical Analysis 1: Comparison: Apligraf vs Control; Test type: Superiority or Other; p = 0.3783, Fisher Exact

4. Secondary Outcome: Degree of Recurrence (Scar Firmness)
Description: Scar firmness measured by Cutometer in millimeters.
Time Frame: Week 52 or Last Visit
Population: mITT population (randomized subjects only). Last Visit is the score recorded at last subject visit with non-missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
mm | 0.2 (0.1) | 0.2 (0.1)
Statistical Analysis 1: Comparison: Apligraf vs Control; Treatment differences in scar firmness evaluated using a 2-tailed Wilcoxon rank sum test with pooled variances; Test type: Superiority or Other; p = 0.7149, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Degree of Recurrence (Scar Thickness)
Description: Scar thickness measured by slide caliper in millimeters. A value of 0.0 mm on the slide caliper is equivalent to normal, non-hypertrophic/raised skin.
Time Frame: Week 52 or Last visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | A (Apligraf) | B (Control)
Number analyzed (Participants) | 12 | 13
mm | 2.0 (2.2) | 1.0 (1.1)
Statistical Analysis 1: Comparison: A (Apligraf) vs B (Control); Treatment differences in scar thickness evaluated using a 2-tailed Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.1670, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Physician Global Assessment
Description: Investigator assessed using 5 point scale (1-excellent, 2-very good, 3-good, 4-moderate, 5-poor)
Time Frame: Week 52 or Last Visit
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
Participants
  Excellent | 3 | 3
  Very Good | 3 | 3
  Good | 0 | 2
  Moderate | 5 | 4
  Poor | 1 | 1
Statistical Analysis 1: Comparison: Apligraf vs Control; Global assessments analyzed as ordinal ranks. Treatment differences in global assessment evaluated using a 2-tailed Wilcoxon rank sum test with pooled variances; Test type: Superiority or Other; p = 0.7221, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Subject Global Assessment
Description: Subject assessed using 5 point scale (1-excellent, 2-very good, 3-good, 4-moderate, 5-poor)
Time Frame: Week 52 or Last Visit
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
Participants
  Excellent | 4 | 6
  Very Good | 1 | 3
  Good | 5 | 2
  Moderate | 2 | 1
  Poor | 0 | 1
Statistical Analysis 1: Comparison: Apligraf vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.4080, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Decreased Utilization of Intralesional Steroid Intervention
Description: The mean number of Intralesional (IL) Injections per participant is reported. A lower number of injections is a better outcome.
Time Frame: 52 weeks
Population: mITT population (randomized subjects only)
Measure: Mean (Standard Deviation); unit: Injections per Participant
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 12 | 13
Injections per Participant | 4.0 (1.8) | 4.2 (1.0)
Statistical Analysis 1: Comparison: Apligraf vs Control; Differences evaluated using a 2-tailed Wilcoxon rank sum test with pooled variances; Test type: Superiority or Other; p = 0.9556, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Apligraf | Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 12/17 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apligraf (N=17) | Control (N=13)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis Viral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Tinea Versicolour (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection Bacterial (Infections and infestations) | 0 (0) | 1 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound Complication (Injury, poisoning and procedural complications) | 5 (8) | 7 (9)
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Vomiting in Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days